CLINICAL TRIAL: NCT07229898
Title: A Phase Ⅰ Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of GEN-725 Tablets in Patients With Advanced Solid Tumors
Brief Title: A Phase Ⅰ Clinical Study of GEN-725 Tablets in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEN-725-R001
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; GEN-725

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Dose-escalation part and dose-expansion part
  Interventions: Drug: GEN-725 tablets

INTERVENTIONS:
Drug: GEN-725 tablets — Dose-escalation part: Subjects received GEN-725 tablets at doses of 4, 6 and 8 mg. A single oral dose was administered on Cycle 1 Day 1, observation was conducted for 4 days (i.e., after oral administration of 1 GEN-725 tablet followed by a 4-day washout period), then once daily from Day 5 onward. Dosing occurred with 21 days of continuous treatment per cycle (from Day 5 to Day 25).
  Dose-expansion part: Subjects received GEN-725 tablets orally at a dose that depends on the outcome of dose-escalation, administered once daily for 21 consecutive days per cycle.

SUMMARY:
A phase Ⅰ clinical study evaluating the safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy of GEN-725 tablets in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form (ICF).
2. Aged ≥ 18 years and ≤ 75 years, regardless of gender.
3. Subjects must meet the following criteria:

   a) Diagnosed by histology or cytology with advanced solid tumors that have progressed after standard treatment, are intolerant to standard treatment, have no standard treatment available, or are judged by the investigator as unsuitable for standard treatment. Tumor types include but are not limited to: NSCLC, HCC, CRC, bladder cancer, breast cancer, etc.; AND b) Time since prior anti-PD-1/PD-L1 monoclonal antibody monotherapy or combination therapy to recurrence/progression is ≥ 6 months.
4. Presence of at least one measurable lesion (RECIST v1.1 criteria).
5. ECOG performance status score of 0 or 1.
6. For HCC patients, must have Child-Pugh class A or B, without hepatic encephalopathy.
7. Expected survival time ≥ 3 months.
8. Toxicities from prior treatments (except for alopecia and pigmentation) have all recovered to Grade 1 or normal levels.
9. Adequate organ function, meeting all of the following laboratory test results prior to enrollment:

   * Hematology: ANC ≥ 1.5×10^9/L, platelet count ≥ 75×10^9/L, hemoglobin ≥ 90 g/L;
   * Liver function: Serum bilirubin ≤ 1.5×upper limit of normal (ULN), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5×ULN, or if liver metastases are present, AST and ALT ≤ 5×ULN;
   * Renal function: Serum creatinine (Cr) ≤ 1.5×ULN, Creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 60 mL/min;
   * Coagulation function: International normalized ratio (INR) ≤ 1.5, Activated partial thromboplastin time (APTT) ≤ 1.5×ULN;
   * Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%.
10. Subjects with reproductive potential (including spouses of male subjects) have no plan for pregnancy or sperm donation from screening until 6 months after the last dose, and are willing to use at least one effective contraception method.

Exclusion Criteria:

1. Subjects with a history of allergic reactions to GEN-725 tablets or to active or inactive excipients of drugs with similar chemical structures or of the same class.
2. Subjects who meet any of the following criteria:

   Have received systemic anti-tumor therapy (including chemotherapy, immunotherapy, biological agents, etc.) within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of the investigational drug;

   Have received hormonal anti-tumor therapy, small molecule targeted therapy, oral fluorouracil drugs, or endocrine therapy within 2 weeks prior to the first dose of the investigational drug;

   Have undergone palliative local therapy for non-target lesions within 2 weeks prior to the first dose of the investigational drug;

   Have received non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, tumor necrosis factor, etc.) within 4 weeks prior to the first dose of the investigational drug;

   Have received Chinese herbal medicines or proprietary Chinese medicines with anti-tumor indications within 2 weeks prior to the first dose of the investigational drug.
3. Subjects who have received anti-tumor vaccines or live vaccines within 4 weeks prior to the first dose of the investigational drug, or who plan to receive such vaccines during the study period.
4. Subjects who have received systemic therapy with corticosteroids (> 10 mg/day of dexamethasone or equivalent dose) or other immunosuppressive drugs within 4 weeks prior to the first dose of the investigational drug. However, topical applications (e.g., ointments, eye drops, inhalants, or nasal sprays) are permitted, provided the dosage does not exceed the recommended dose in the prescribing information and there are no signs of systemic exposure.
5. Subjects with a history of acute or chronic pancreatitis.
6. Subjects with brain metastases and/or carcinomatous meningitis (except for those with brain metastases that have been adequately treated, have remained stable for at least 3 months prior to screening, have all neurological symptoms returned to baseline levels, show no evidence of new or enlarging metastases, and have ceased radiotherapy, surgery, or steroid therapy for at least 4 weeks prior to the first dose of the investigational drug).
7. Subjects with spinal cord compression that has not been radically treated by surgery and/or radiotherapy.
8. Subjects with a history or evidence of significant cardiovascular disease within 6 months prior to screening, including but not limited to:

   History of myocardial infarction, coronary angioplasty or bypass grafting, valvular heart disease or valvular repair, clinically significant arrhythmias requiring treatment, unstable angina, transient ischemic attack, cerebrovascular accident, etc.;

   Congestive heart failure classified as Class III or IV according to the New York Heart Association (NYHA) criteria.
9. Subjects with clinically significant abnormalities in the 12-ECG examination during screening, including but not limited to severe arrhythmias, prolonged QT interval (QTcF: > 450 ms for males, > 470 ms for females; QTc interval calculated using Fridericia's formula); or the presence of any condition that may increase the risk of QT prolongation, such as a known history of QTc prolongation, congenital long QT syndrome, Brugada syndrome, torsades de pointes, uncontrolled electrolyte disturbances (e.g., hypocalcemia, hypokalemia, hypomagnesemia, etc.).
10. Subjects with hypertension uncontrolled by antihypertensive medication (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg).
11. Subjects with presence of persistent or active infection that remains poorly controlled despite medication, including but not limited to:

    Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus (HBV) deoxyribonucleic acid (DNA) quantification ≥ the upper limit of normal (ULN);

    Hepatitis C virus antibody (HCV-Ab) positive and hepatitis C virus (HCV) ribonucleic acid (RNA) ≥ ULN;

    Note: HBV-DNA testing is required only for HBsAg positive subjects; HCV-RNA testing is required only for HCV-Ab positive subjects.
12. Subjects with existing autoimmune diseases or related symptoms, or a history of autoimmune diseases, immunodeficiency diseases (e.g., leukemia, HIV, etc.), or a history of organ transplantation.
13. Subjects with active, uncontrolled systemic infection (e.g., bacterial, viral, or fungal) despite optimal therapy.
14. Subjects with a history of or current interstitial lung disease, pulmonary fibrosis, drug-induced interstitial pneumonia, or radiation pneumonitis requiring steroid treatment.
15. Subjects with moderate to large pleural effusion, pericardial effusion, or ascites requiring pharmacological or medical intervention.
16. Subjects who have had other malignancies ( except radically cured basal cell carcinoma of the skin, squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix, etc.) within 5 years prior to the first dose of the investigational drug, except for the tumor being treated in this study.
17. Subjects who have undergone major surgery within 3 months prior to screening and have not fully recovered, or who plan to undergo major surgery during participation in this study (except for outpatient surgeries judged by the investigator to have no impact on subject safety or trial outcomes).
18. Subjects with uncontrollable nausea, vomiting, inability to swallow normally, or those with chronic gastrointestinal diseases, gastrointestinal obstruction, or other conditions that may affect the administration and absorption of the investigational drug.
19. Subjects with a documented history of psychiatric disorders, or a history of psychotropic drug abuse, drug abuse, or alcohol abuse.
20. Women who are pregnant or breastfeeding.
21. Subjects who have participated in any other drug clinical trial or are receiving other investigational therapies within 4 weeks prior to the first dose of the investigational drug (or within 5 half-lives of another investigational drug, whichever is longer) (except for patients participating only in the overall survival follow-up phase of a study).
22. Any other condition deemed by the investigator as inappropriate for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Dose-Limiting Toxicity (DLT) (Dose-escalation part) | Day 25
Incidence and severity of adverse events (AEs) (Dose-escalation part) | From the signing of the Informed Consent Form (ICF) by the subjects until 28±7 days after the last administration of the study drug.
  AEs are assessed based on NCI CTCAE v5.0.
Overall Response Rate (ORR) (Dose-expansion part) | Up to approximately 24 months.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of GEN-725 (Dose-escalation part and dose-expansion part) | Up to 72 hours post-dose in dose-escalation part and 24 hours post-dose in dose-expansion part.
Time to Maximum Plasma Concentration (Tmax) of GEN-725 (Dose-escalation part and dose-expansion part) | Up to 72 hours post-dose in dose-escalation part and 24 hours post-dose in dose-expansion part.
Steady-State Valley Concentration (Css,min) of GEN-725 (Dose-escalation part and dose-expansion part) | Up to Day 26 in dose-escalation part and Day 22 in dose-expansion part.
Steady-State Peak Concentration (Css,max) of GEN-725 (Dose-escalation part and dose-expansion part) | Up to Day 26 in dose-escalation part and Day 22 in dose-expansion part.
Overall Response Rate (ORR) (Dose-escalation part) | Up to approximately 24 months.
Disease Control Rate (DCR) (Dose-escalation part and dose-expansion part) | Up to approximately 24 months.
Duration of Response (DOR) (Dose-escalation part and dose-expansion part) | Up to approximately 24 months.
Progression-Free Survival (PFS) (Dose-escalation part and dose-expansion part) | Up to approximately 24 months.
Overall Survival (OS) (Dose-escalation part and dose-expansion part) | Up to approximately 24 months.
Evaluation of life quality per EORTC QLQ-C30 score changes (Dose-escalation part and dose-expansion part) | Up to approximately 24 months.
Incidence and severity of adverse events (AEs) (Dose-expansion part) | From the signing of the Informed Consent Form (ICF) by the subjects until 28±7 days after the last administration of the study drug.
  AEs are assessed based on NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Harbin Medical University Cancer Hospital, Harbin
  - Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute, Shandong Cancer Hospital), Jinan
  - Shanghai East Hospital, Shanghai
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang